CLINICAL TRIAL: NCT06692569
Title: The Effect of Modified Constraint Induced Movement Therapy on Upper Extremity Function in Stroke Rehabilitation
Acronym: mCIMT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Collaborators: Majmaah University (Other)
Responsible Party: Principal Investigator, Karthick Balasubramanian, Lecturer, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUREC-May.22/COM-2022/6-1
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Hemiplegia; Chronic Stroke Patients
Keywords: stroke; hemiplegia; constraint induced movement therapy; modified constraint induced movement therapy; trunk restrain; upper extremity motor function
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Conventional Physical Therapy
  Interventions: Other: Conventional Physical Therapy
- Experimental (Experimental): Conventional Physical Therapy and modified constraint induced movement therapy
  Interventions: Other: Modified Constraint Induced Movement Therapy

INTERVENTIONS:
Other: Conventional Physical Therapy — The conventional Physical Therapy, the treatment will be based on the client's capabilities. It included functional reeducation, muscle strengthening and stretching, muscle tone regulation methods, and training for activities of daily living
  Arms: Control
Other: Modified Constraint Induced Movement Therapy — Modified Constraint Induced Movement Therapy (mCIMT) which involves trunk constraint along with conventional Physical Therapy treatment. Under the attentive guidance of a physiotherapist, the patient engages in specific hand activities aligned with personalized goals. These activities encompass tasks such as picking up marbles, flipping cards, stacking blocks, combing hair, writing, and other actions relevant to daily life. The difficulty level is dynamically adjusted according to the patient's abilities and progress during the training sessions.Tasks may vary from one patient to another, and each session introduces fresh, goal-oriented challenges to further enhance rehabilitation outcomes, along with the conventional physical therapy treatment. The patients were wearing a trunk west which had a Velcro strap on the non-effected side part of the west, and it was attached to the Velcro straps on the non-affected part on the back support of the treatment chair.
  Arms: Experimental

SUMMARY:
The purpose of the study is to determine the effect of Modified Constraint-Induced Movement Therapy and trunk restraint contrasted with conventional physical therapy treatment on improving upper extremity function, balance, and quality of life among chronic hemiplegic patients.

* To find out the effectiveness of conventional physical therapy treatment on improving upper extremity function, balance, and quality of life among chronic hemiplegic patients.
* To find out the effectiveness of modified constraint induced movement therapy (mCIMT) and trunk restraint along with conventional physical therapy treatment on improving upper extremity function, balance, and quality of life among chronic hemiplegic patients.
* To find out the effectiveness of modified constraint induced movement therapy (mCIMT) and trunk restraint combined with conventional physical therapy treatment versus conventional physical therapy treatment alone on improving upper extremity function, balance, and quality of life among chronic hemiplegic patients.

ELIGIBILITY:
Inclusion Criteria:

* Right or left-sided chronic hemiplegic patients.
* Onset of stroke More than six months.
* Age between 45 to 65 years of both genders.
* Mini-Mental State Examination - Scored more than 24/30.
* Modified Ashworth Scale for spasticity 1 or 1+.
* Have at least 20° wrist active extension and at least 10° of metacarpophalangeal active extension of the paretic upper extremity.
* Have at least grade 2/5 of muscle power on upper extremity especially in wrist extensors.
* Have normal visual perception.
* With no other neurological disorders.

Exclusion Criteria:

* Unable to follow visual and oral commands.
* Unilateral neglect.
* Severe cognitive, or language deficits.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-07-13 (Estimated); Study Completion 2025-07-13 (Estimated)

PRIMARY OUTCOMES:
Wolf Motor Function Test | Week 0 and week 6
  Wolf Motor Function Test assessment tool was specifically developed to assess and evaluate the exercise capacity of individuals with varying degrees of upper extremity motion impairments, ranging from mild to severe, in both laboratory and clinical settings. It represents an enhancement over a previous tool that was more suitable for assessing high-functioning patients but posed challenges when used with individuals who had limited hand and finger mobility
Berg Balance Scale | week 0 and week 6
  The Berg Balance Scale (BBS) is a widely used clinical assessment tool designed to evaluate and quantify an individual's balance and stability during various tasks. It consists of a series of 14 tasks or activities that challenge balance and mobility, such as standing on one foot, reaching for objects, and turning in place. Each task is scored on a scale ranging from 0 to 4, with 0 indicating the lowest level of performance and 4 indicating the highest level of performance
Stroke Specific Quality of Life Scale | week 0 and week 6
  Stroke Specific Quality of Life Scale (SS-QOL) is a specialized assessment tool designed to measure the quality of life in individuals who have experienced a stroke. This scale is specifically tailored to evaluate the impact of stroke on various aspects of a person's life, encompassing physical, psychological, and social domains. The SS-QOL questionnaire typically consists of multiple items or questions that cover a range of topics, including physical health, mobility, communication abilities, emotional well-being, and social relationships. Respondents rate their level of satisfaction or well-being in each domain, often on a scale from 0 to 5 or 0 to 100, with higher scores indicating better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Karthick BALASUBRAMANIAN, MPT, Principal Investigator — University of Jazan
Locations (1):
- Majmaah Rehabilitation center, Riyadh, Riyadh Region, Saudi Arabia

REFERENCES:
- [Derived] M Shahhar A, Shaik AR, Esht V, Alshehri MM, Balasubramanian K, Ramasamy Sanjeevi R, Abdulrahman Alfaleh K, Okab Alsalem W, Fathi WA, A Alothman S. Modified Constraint-Induced Movement Therapy with Trunk Restraint for Upper Extremity Functional Motor Recovery, Balance and Health-Related Quality of Life in Chronic Stroke: A Single-Blinded Randomized Controlled Clinical Trial. NeuroRehabilitation. 2026 Feb 2:10538135261417372. doi: 10.1177/10538135261417372. Online ahead of print. PMID 41627128